CLINICAL TRIAL: NCT06339879
Title: Health Effects of Grain Foods in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Grain Foods Foundation (Unknown)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-2023-1071
Record Dates: First submitted 2023-12-11; First posted 2024-04-01 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: High Whole Grain and Low Sugar; Medium Whole Grain and Low Sugar; Low Whole Grain and Low Sugar; Low Whole Grain and High Sugar
Keywords: whole grain; refined grain; glycemia; appetite; food intake; microbiome; body weight; blood pressure; lipemia; hedonics
MeSH Terms: conditions — Body Weight; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High Whole Grain, Low Sugar (Active Comparator): 6 servings of whole grain and <13% energy from added sugars.
  Interventions: Other: High Whole Grain, Low Sugar
- Low Whole Grain, Low Sugar (Active Comparator): 3 servings of whole grain and <13% energy from added sugars.
  Interventions: Other: Low Whole Grain, Low Sugar
- High Whole Grain, High Sugar (Active Comparator): 6 servings of whole grain and >13% energy from added sugars.
  Interventions: Other: High Whole Grain, High Sugar
- Low Whole Grain, High Sugar (Active Comparator): 3 servings of whole grain and >13% energy from added sugars.
  Interventions: Other: Low Whole Grain, High Sugar

INTERVENTIONS:
Other: High Whole Grain, Low Sugar — 6 servings of whole grain and <13% energy from added sugars.
  Arms: High Whole Grain, Low Sugar
Other: Low Whole Grain, Low Sugar — 3 servings of whole grain and <13% energy from added sugars.
  Arms: Low Whole Grain, Low Sugar
Other: High Whole Grain, High Sugar — 6 servings of whole grain and >13% energy from added sugars.
  Arms: High Whole Grain, High Sugar
Other: Low Whole Grain, High Sugar — 3 servings of whole grain and >13% energy from added sugars.
  Arms: Low Whole Grain, High Sugar

SUMMARY:
This study will assess the effects of eating whole grain foods versus refined grain foods with different amounts of added sugar. It is hypothesized that a diet including grain products will have beneficial effects on taste hedonics, appetite, food/energy intake, body weight, blood pressure, acute and chronic glycemia and acute and chronic lipemia compared to customary diets controlling for added sugars, saturated fats and sodium.

DETAILED DESCRIPTION:
This 16-week, randomized, controlled, parallel-arm, clinical trial will assess the effects of consuming four different categories of grain foods on taste hedonics, appetite, food/energy intake, body weight, and blood pressure as well as acute and longer-term glycemia and lipemia. It will also examine the effects of foods varying in grain/carbohydrate composition on the microbiome and microbiota functionality. One hundred and twenty adults will be recruited and randomly assigned to one of four intervention groups. These groups will be defined by the diets they are prescribed. All will be prescribed diets containing approximately 50%; 35% and 15% energy from carbohydrate, fat and protein, respectively. Grain foods will comprise 50% of the carbohydrate component (i.e., 25% of total energy). The grain foods will be assigned to one of four categories based on whole grain content and concentrations of added sugars. The grain foods meeting these criteria will have the following composition:

Group 1 - High Whole Grain, Low Sugar 6 servings of whole grain and <13% energy from added sugars.

Group 2 - Low Whole Grain, Low Sugar 3 servings of whole grain and <13% energy from added sugars.

Group 3 - High Whole Grain, High Sugar 6 servings of whole grain and >13% energy from added sugars.

Group 4 - Low Whole Grain, High Sugar 3 servings of whole grain and >13% energy from added sugars.

Detailed Study Design

The study measures and timing are outlined in the following table:

Screening Week 1 Baseline Week 2 Week 5 Week 8 Week 11 Week 14 Fasting Blood X X X XX MTT X X X Weight X X X X X X Body Composition X X CGM X X X Intake X Hedonics (palatability) X X X Appetite X X X Activity X X X Blood Pressure X X X X X X Microbiota X X X X X Compliance X X X X X MTT = Meal Tolerance Test; DXA= Dual-energy X-ray Absorptiometry; CGM=Continuous glucose monitoring

ELIGIBILITY:
Inclusion Criteria:

* male and female; 21 to 60 years old; Hemoglobin A1c concentration between 5.7 and 6.4%
* Prefer no use of medications, but if on medication, must have been on a stable dose for 3 months and plan to remain at the same dose for the duration of the trial.
* low customary intake of whole grain foods (less than 2 servings per day) and high energy from added sugar (greater than 10% energy).

Exclusion Criteria:

* Grain or dairy sensitivities or allergies or celiac disease; sensitivity or allergy to other foods that would result in refusal to eat a class of foods.
* smoker
* intended weight loss or gain during the study period; intended change of activity level during the study period
* use of blood thinners
* prior gastrointestinal surgery.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemia | 12 weeks
  blood sugar

SECONDARY OUTCOMES:
Appetite | 12 weeks
  ingestive sensations measured by VAS ratings scale 1 (lowest) - 100 (highest)
Taste Hedonics | 12 weeks
  palatability
Energy Intake | 12 weeks
  kcals
Body Weight | 12 weeks
  pounds
Systolic and Diastolic Blood Pressure | 12 weeks
  mm mercury
Lipemia | 12 weeks
  Blood lipids

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
deidentified data will be shared.